CLINICAL TRIAL: NCT00659815
Title: Performance of Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution in a Clear Polyethylene Terephthalate (PET) Bottle.
Brief Title: Performance of Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution in a New Packaging Configuration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 549
Record Dates: First submitted 2008-04-12; First posted 2008-04-16 (Estimated); Results first posted 2010-11-15 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Comfort

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReNu in Currently Marketed Bottle (Active Comparator): Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution Packaged in the Currently Marketed Resin Bottle.
  Interventions: Device: Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution Packaged in the Currently Marketed Resin Bottle.
- ReNu in Clear Resin Bottle (Experimental): Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution Packaged in a Clear Resin Bottle.
  Interventions: Device: Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution Packaged in a Clear Resin Bottle.

INTERVENTIONS:
Device: Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution Packaged in the Currently Marketed Resin Bottle. — Daily care for contact lenses.
  Arms: ReNu in Currently Marketed Bottle
Device: Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution Packaged in a Clear Resin Bottle. — Daily care for contact lenses
  Arms: ReNu in Clear Resin Bottle

SUMMARY:
The objective of the study is to evaluate the product performance of Bausch & Lomb ReNu MultiPlus Multi-Purpose Solution in a new packaging configuration

ELIGIBILITY:
Inclusion Criteria:

* Subject is a habitual wearer of planned replacement soft contact lenses
* VA correctable to 0.3 LogMar or better (driving vision)
* Clear central cornea
* Subject uses a lens care system on a regular basis

Exclusion Criteria:

* Systemic disease affecting ocular health
* Using systemic or topical medications
* Wear monovision, multifocal or toric contact lenses
* Any grade 2 or greater slit lamp findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Cairns, PhD, MCOptom, Study Director — Bausch & Lomb Incorporated; James Ferrari, OD, Principal Investigator — James Ferrari, OD
Locations (1):
- James Ferrari, OD, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 23 investigative sites in the United States. First participant was enrolled 3/19/2008, last participant exited the study 5/19/08.
Pre-assignment Details: 312 Participants were enrolled, 2 participants were ineligible at baseline but were dispensed lens care solution and completed the study. 2 participants were not dispensed lens care solution. 308 eligible subjects started the study, 8 were discontinued during the study. 300 participants completed the study.
Groups:
- Marketed Bottle ReNu MultiPlus Multi-Purpose Solution: Currently Marketed high-density polyethylene (HDPE) Bottle with B&L ReNu MultiPlus Multi-Purpose Solution for 1 month, daily contact lens care.
- Clear Bottle ReNu MultiPlus Multi-Purpose Solution: Clear polyethylene terephthalate (PET) Bottle with B&L ReNu MultiPlus Multi-Purpose Solution for 1 month daily contact lens care.
Period: Overall Study
Arm/Group | Marketed Bottle ReNu MultiPlus Multi-Purpose Solution | Clear Bottle ReNu MultiPlus Multi-Purpose Solution
Started | 157 | 151
Completed | 153 | 147
Not Completed | 4 | 4
Not completed — Study related symptoms and complaints | 2 | 1
Not completed — Inability to maintain wearing schedule | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marketed Bottle ReNu MultiPlus Multi-Purpose Solution | Clear Bottle ReNu MultiPlus Multi-Purpose Solution | Total
Number analyzed (Participants) | 157 | 151 | 308
Age, Customized [Number; unit: Participants]
  >=18 and <=65 years | 157 | 151 | 308
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 111 | 230
  Male | 38 | 40 | 78
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 3 | 6 | 9
  White | 144 | 136 | 280
Region of Enrollment [Number; unit: participants]
  United States | 157 | 151 | 308

OUTCOME MEASURES:

1. Primary Outcome: Comfort
Description: Non-inferiority assessment of symptoms/complaints to rate solution comfort. Measurement based on 0-100 scale for each eye. Zero represented the least favorable rating and 100 represented the most favorable rating.
Time Frame: Over-all follow-up visits from baseline to 1 month
Population: Symptoms/Complaints Over-All Scheduled Follow-Up Visits (All Eligible, Dispensed Eyes with non-missing scores)
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: eyes
Arm/Group | Marketed Bottle ReNu MultiPlus Multi-Purpose Solution | Clear Bottle ReNu MultiPlus Multi-Purpose Solution
Number analyzed (Participants) | 156 | 150
Number analyzed (eyes) | 312 | 300
Units on a Scale
  Comfort | 90.2 (12.7) | 92.7 (9.3)
  End of Day Comfort | 84.5 (16.9) | 87.2 (14.5)
  Burning/Stinging on Insertion | 90.3 (15.8) | 93.2 (13.9)
  Irritation | 90.2 (14.1) | 92.9 (10.6)
  Itching | 93.0 (10.7) | 94.9 (9.3)
  Dryness | 88.8 (14.4) | 90.5 (11.8)
  Redness | 93.4 (11.8) | 94.0 (11.2)
  Vision | 93.5 (12.4) | 95.7 (7.8)
  Lens Cleanliness | 92.7 (12.4) | 92.7 (12.4)
  Lens Handling | 96.7 (7.3) | 95.3 (10.3)

2. Primary Outcome: Slit Lamp Findings
Description: Graded 0-4 where Grade 0=none; Grade 1=Trace; Grade 2=Mild; Grade 3=Moderate; Grade 4=Severe.
Time Frame: Over-all follow-up visits from baseline to1 month
Population: Graded Slit Lamp Findings over All Follow-Up Visits (Any finding, All Dispensed Eyes, 151 + 2 possible).
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | Marketed Bottle ReNu MultiPlus Multi-Purpose Solution | Clear Bottle ReNu MultiPlus Multi-Purpose Solution
Number analyzed (Participants) | 156 | 152
Number analyzed (eyes) | 312 | 304
Eyes
  Slit Lamp Finding > Grade 2 | 1 | 0
  Slit Lamp Findings </= Grade 2 | 311 | 304

3. Primary Outcome: Lens Deposits
Description: Lens Deposits (All Eligible, Dispensed Eyes) Absent = deposit ratings of none or light; Present = deposit ratings of medium or heavy.
Time Frame: Over-all study visits, baseline to 1-month
Population: Lens deposits over all scheduled follow-up visits (all eligible, dispensed eyes with non-missing data)
Measure: Number; unit: Eyes
Units Other Than Participants: eyes
Arm/Group | Marketed Bottle ReNu MultiPlus Multi-Purpose Solution | Clear Bottle ReNu MultiPlus Multi-Purpose Solution
Number analyzed (Participants) | 155 | 150
Number analyzed (eyes) | 310 | 300
Eyes
  Absent | 292 | 281
  Present | 18 | 19

ADVERSE EVENTS:
Time Frame: One month
Arm/Group | Marketed Bottle ReNu MultiPlus Multi-Purpose Solution | Clear Bottle ReNu MultiPlus Multi-Purpose Solution
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/151
Other Adverse Events (participants affected / at risk) | 0/157 | 0/151

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the investigator(s) after the review by, and in consultation and agreement with the Sponser, and such that confidential or proprietary information is not disclosed.